CLINICAL TRIAL: NCT05063526
Title: The Role of Diaphragmatic Ultrasound as a Predictor of Successful Extubation From Mechanical Ventilation in Respiratory Intensive Care Unit
Brief Title: The Role of Diaphragmatic Ultrasound as a Predictor of Extubation From Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ahmed Aelgharib Ahmed, Principal Investigator, Beni-Suef University
Other Study IDs: FMBSUREC/05012020/Ahmed
Record Dates: First submitted 2021-09-03; First posted 2021-10-01 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Diaphragm Ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group B: 40 patients who are mechanically ventilated due to pulmonary disease at respiratory ICU had their diagnosis as follows: 21 (53%) had COPD, 8 (20%) had asthma, 5 (13%) had bronchiectasis, 5 (13%) had pneumonia and
  1 (3%) had viral influenza H1N1. Out of group B patients, 11 patients (13.75%) had failed weaning, of which 6 patients needed reintubation and 5 patients needed non-invasive positive ventilation of which 3 patients were re-intubated and 2 patients died.
  Interventions: Device: ultrasound
- Group A: 40 patients on mechanical ventilation due to non-pulmonary disease at respiratory ICU had their diagnosis as follows: 24 (60%) had congestive heart failure, 4 (10%) had diabetes mellitus, 4 (10%) had sepsis other than pneumonia, 2 (5%) had epilepsy, 2 (5%) had embolic hemiplegia, and 4 (10%) had chronic renal failure. Out of group A patient, 9 patients (11.25%) had failed weaning of which 4 patients needed reintubation and 5 patients needed non-invasive positive ventilation of which 2 patients were reintubated and 3 patients died.
  Interventions: Device: ultrasound
- control group.: 40 patients Chronic obstructive pulmonary disease (COPD) from Outpatient Clinic
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — ultrasound on diaphragm

SUMMARY:
Aim: To evaluate real-time ultrasound in the evaluation of diaphragmatic thickening, thickening fraction and or excursion to predict extubation outcomes. The investigators aimed to compare these parameters with other traditional weaning measures.

DETAILED DESCRIPTION:
The diaphragm is an important respiratory muscle and dysfunction is very common in patients receiving mechanical ventilation. Diaphragm fatigue occurs even in patients who successfully pass the Spontaneous Breathing Test (SBT). Interrupting ventilation too early can lead to increased cardiovascular and respiratory pressure (CO2).retention and hypoxemia with up to 25% of patients requiring reinstitution of ventilator support. Unnecessary delays in liberation from mechanical ventilation also can be deleterious. Complications such as ventilator-associated pneumonia and ventilator-induced diaphragm atrophy can be seen with short periods of mechanical ventilation thereby prolonging mechanical ventilation. As SBT monitoring is insensitive to detect early signs of load-capacity imbalance. The evaluation of the diaphragmatic thickening fraction (DTF) may be also helpful to assess diaphragmatic function and its contribution to respiratory workload. Ultrasound can be used to detect the deflection of the diaphragm, which helps to identify patients with diaphragm dysfunction

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients intubated for more than 48 hours who are ready for weaning with the following criteria.

  1. positive end-expiratory pressure (PEEP) ≤ 5 cm H2O.
  2. Fraction of inspired oxygen (FiO2) < 0.5.
  3. respiratory rate (RR) < 30 breaths/min.
  4. rapid shallow breathing index < 105, PaO2/FiO2 > 200.
* Age< 65 years.

Exclusion Criteria:

* Age<18 years.
* Patient with history of plural effusion, trauma to chest and history of mechanical ventilation for < 6 months.
* patient with neuromuscular diseases affect diaphragm .

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This prospective study was carried out on 40 patients who are mechanically ventilated due to pulmonary disease, 40 patients on mechanical ventilation due to non-pulmonary disease at respiratory ICU and 40Chronic obstructive pulmonary disease (COPD) patients from Outpatient Clinic serving as controls at Embaba Chest Hospital. Cairo, Egypt during a period from January 2018 to November 2019. Written informed consent was obtained from all patients prior to enrollment according to approval at the local committee of Beni-suef University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
diaphragmatic ultrasound thickening | during weaning from mechanical ventilation 0n T- tube, through study completion, an average of 1 year
  Right diaphragmatic ultrasound measurement thickening in millimeter was made during tidal and deep breathing . patient is in the supine position and measurement of right diaphragm by M-mode and B-mode images
diaphragmatic ultrasound thickening fraction | during weaning from mechanical ventilation 0n T- tube, through study completion, an average of 1 year
  Right diaphragmatic ultrasound measurement thickening fraction(percentage% ) was made during tidal and deep breathing . patient is in the supine position and measurement of right diaphragm by M-mode and B-mode images
diaphragmatic ultrasound excursion | during weaning from mechanical ventilation 0n T- tube, through study completion, an average of 1 year
  Right diaphragmatic ultrasound measurement excursion( centimeter) was made during tidal and deep breathing . patient is in the supine position and measurement of right diaphragm by M-mode and B-mode images

SECONDARY OUTCOMES:
diaphragmatic ultrasound thickening fraction | Up to 48 hours on T-tube, through study completion, an average of 1 year
  Differences in thickening fraction ( millimeter )between patients who are successfully and failed weaning .
diaphragmatic ultrasound thickening | Up to 48 hours on T-tube, through study completion, an average of 1 year
  Differences in diaphragm thickening(percentage% )between patients who are successfully and failed weaning .
diaphragmatic ultrasound excursion | Up to 48 hours on T-tube, through study completion, an average of 1 year
  Differences in diaphragm excursion ( centimeter) between patients who are successfully and failed weaning

CONTACTS AND LOCATIONS:
Overall Officials: Randa S Mohamed, professor, Study Director — Benisuef unviresity
Locations (1):
- Beni-suef, Banī Suwayf, Mequbal, Egypt

REFERENCES:
- [Background] Ferrari G, De Filippi G, Elia F, Panero F, Volpicelli G, Apra F. Diaphragm ultrasound as a new index of discontinuation from mechanical ventilation. Crit Ultrasound J. 2014 Jun 7;6(1):8. doi: 10.1186/2036-7902-6-8. eCollection 2014. PMID 24949192
- [Background] Grosu HB, Lee YI, Lee J, Eden E, Eikermann M, Rose KM. Diaphragm muscle thinning in patients who are mechanically ventilated. Chest. 2012 Dec;142(6):1455-1460. doi: 10.1378/chest.11-1638. PMID 23364680
- [Background] Farghaly S, Hasan AA. Diaphragm ultrasound as a new method to predict extubation outcome in mechanically ventilated patients. Aust Crit Care. 2017 Jan;30(1):37-43. doi: 10.1016/j.aucc.2016.03.004. Epub 2016 Apr 22. PMID 27112953
- [Background] Umbrello M, Formenti P. Ultrasonographic Assessment of Diaphragm Function in Critically Ill Subjects. Respir Care. 2016 Apr;61(4):542-55. doi: 10.4187/respcare.04412. Epub 2016 Jan 26. PMID 26814218